CLINICAL TRIAL: NCT00797186
Title: Less Invasive Detection and Treatment of Very Early Coronary Artery Disease in Patients With Diabetes Mellitus Using Regadenoson Stress Cardiac Magnetic Resonance Imaging
Brief Title: Less Invasive Detection and Treatment of Very Early Coronary Artery Disease in Patients With Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Pfizer (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Angela M. Taylor, MD, University of Virginia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13761; 1K23HL093118-01 (NIH)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Type 2 Diabetes; Microvascular Dysfunction
Keywords: diabetes; dyslipidemia; microvascular dysfunction; imaging
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensive therapy (Other): There is one arm in this trial. All patients receive the same therapy. The goal is to compare a noninvasive and invasive imaging technique in the same population.
  Interventions: Other: Intensive risk factor management

INTERVENTIONS:
Other: Intensive risk factor management — Aggressive medical and lifestyle therapy.

SUMMARY:
This protocol focuses on the development of a noninvasive method of early coronary artery disease detection in diabetes. The overall hypothesis is that risk factors for the metabolic syndrome will predict invasive findings on intravascular ultrasound (IVUS) and noninvasive findings on cardiac magnetic resonance (CMR) perfusion imaging. Secondary objectives will include demonstrating the relative importance of individual risk factors early in disease, demonstrating the positive effects of aggressive risk factor modification on disease, demonstrating the relative importance of treatment of individual risk factors on disease progression or stabilization, and that invasive findings on IVUS will predict noninvasive findings with CMR. Such techniques may allow earlier noninvasive detection of disease as well as tailor treatment early in the disease process making prevention more cost effective.

The specific aims of this proposal are as follows:

1. To assess whether risk factors for coronary artery disease, both known and novel, predict quantitative and qualitative plaque characteristics on IVUS and alterations in myocardial blood flow on CMR.
2. To assess whether improvements in risk factors through aggressive treatment improve microvascular function as measured by CMR and plaque stabilization and/or regression as measured by IVUS.
3. To assess which risk factors are most predictive early in disease and to demonstrate which risk factors, when treated, provide the most benefit.
4. To assess whether findings on CMR predict findings on IVUS, thus, providing a noninvasive method of early disease detection.

DETAILED DESCRIPTION:
Type II Diabetes has become an epidemic in the United States. Cardiovascular disease is the most common cause of death in this population and is two to four fold higher than the general population. This increased risk is at least partially attributable to the high prevalence of the metabolic syndrome with its multiple coronary heart disease risk factors including central obesity, hypertension, glucose intolerance, chronic inflammation, and dyslipidemia. However, recent trials have demonstrated that traditional risk factors alone are not completely predictive of disease burden particularly early in the disease process prior to the development of flow-limiting coronary stenoses. Diagnosis and prevention of cardiovascular disease development has, thus, been elusive in this high risk population. It is not entirely clear which factors, known or novel, contribute the most in very early disease and which therapies may be most beneficial.

It has been suggested that microvascular dysfunction, a composite of endothelial dysfunction, abnormal blood cell rheology, and abnormal blood viscosity, precedes the development of overt coronary stenoses and contributes to increased cardiovascular risk very early in disease development. Microvascular reactivity is affected by many aspects of the metabolic syndrome. Commonly used tools may not be adequate to evaluate microvascular function in the heart at baseline or in response to therapy. Myocardial contrast echocardiography (MCE) and cardiac magnetic resonance imaging (CMR) provide noninvasive technology capable of directly measuring microvascular function within the heart. Our preliminary data with these modalities shows significantly reduced microvascular function in diabetes in the absence of distinct coronary stenoses.

Prior to development of stenoses in the coronary arteries, plaque accumulates via positive remodeling preserving the lumen. This can be detected invasively through the use of intravascular ultrasound (IVUS). Coronary CT is a potential noninvasive modality able to assess this early remodeling process, but it requires a substantial radiation dose and iodinated contrast dye. In addition, CT requires calcification to have occurred within the plaque, a finding believed to occur well into the life of the plaque. It is unclear how early plaque development is related to microvascular function and if stabilization or regression of plaque with available therapies improves microvascular function.

The overall hypothesis is that risk factors for the metabolic syndrome will predict invasive findings on IVUS and noninvasive findings on CMR perfusion imaging. Secondary objectives will include demonstrating the relative importance of individual risk factors early in disease, demonstrating the positive effects of aggressive risk factor modification on disease, demonstrating the relative importance of treatment of individual risk factors on disease progression or stabilization, and that invasive findings on IVUS will predict noninvasive findings with CMR. Such techniques may allow earlier noninvasive detection of disease as well as tailor treatment early in the disease process making prevention more cost effective.

The specific aims of this proposal are as follows:

1. To assess whether risk factors for coronary artery disease, both known and novel, predict quantitative and qualitative plaque characteristics on IVUS and alterations in myocardial blood flow on CMR. This will be accomplished by performing IVUS during cardiac catheterization followed by CMR perfusion imaging in subjects at baseline. Risk factors will be assessed by the following methods: history, physical exam, and laboratory testing. As CMR has the ability to detect global dysfunction, as opposed to current commonly used noninvasive techniques, the hypothesis is that risk factors for cardiovascular disease will predict findings on IVUS as well as CMR.
2. To assess whether improvements in risk factors through aggressive treatment improve microvascular function as measured by CMR and plaque stabilization and/or regression as measured by IVUS. Subjects will be treated aggressively according to current American College of Cardiology and American Diabetes Association recommendations in the Diabetes Cardiovascular Clinic and will be reassessed at one year. The hypothesis is that improvement in risk factors will predict improvements in measurements by IVUS and MRI.
3. To assess which risk factors are most predictive early in disease and to demonstrate which risk factors, when treated, provide the most benefit. As the metabolic syndrome is present for as many as 10 years prior to the development of diabetes, the hypothesis is that risk factors associated directly with the metabolic syndrome will be most predictive of disease and disease improvement.
4. To assess whether findings on CMR predict findings on IVUS, thus, providing a noninvasive method of early disease detection. The hypothesis is that MRI will predict findings on IVUS, providing a novel noninvasive mechanism for direct detection of early coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Metabolic Syndrome
* Not all risk factors at goal
* Willingness to attend frequent clinic visits
* No coronary stenosis greater than 50% found on catheterization

Exclusion Criteria:

* Type 1 diabetes
* GFR less than 60ml/min/1.73m2
* Females who are pregnant, lactating, not using reliable contraceptive method
* Known coronary stenosis greater than 50%
* Subjects in which stress testing would be contraindicated
* Prior heart transplantation
* Expected survival less than one year
* HIV infection
* Hepatorenal syndrome or history of liver transplant
* Contraindication to MRI
* Significant pulmonary hypertension

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
LDL density | 1 year
HDL | 1 year
change in microvascular perfusion | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States